CLINICAL TRIAL: NCT01889758
Title: Pharmacokinetic Studies of Tacrolimus in Transplant Patients
Acronym: PK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: University of Colorado, Denver (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Rita Alloway, Research Professor of Medicine, University of Cincinnati
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: U01 Grant; FDA UO1 Grant (Other Grant/Funding Number: 1UO1FD004573)
Record Dates: First submitted 2013-06-21; First posted 2013-06-28 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Kidney Transplant Recipients; Liver Transplant Recipients
Keywords: bioequivalence; tacrolimus; kidney; liver; transplant
MeSH Terms: interventions — Tacrolimus; lepirudin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sequence 1 (Active Comparator): Tacrolimus Hi for 1 week with full PK on Day 7, then tacrolimus Lo for 1 week with full PK on Day 14, then Prograf for 1 week with full PK on Day 21, then tacrolimus Hi with full PK on Day 28, then Prograf for 1 week with full PK on Day 35, and then tacrolimus Lo for 1 week with full PK on Day 42
  Interventions: Drug: Prograf; Drug: Tacrolimus
- Sequence 2 (Active Comparator): Tacrolimus Lo for 1 week with full PK on Day 7, then Prograf for 1 week with full PK on Day 14, then tacrolimus Hi for 1 week with full PK on Day 21, then tacrolimus Lo with full PK on Day 28, then tacrolimus Hi for 1 week with full PK on Day 35, and then Prograf for 1 week with full PK on Day 42
  Interventions: Drug: Prograf; Drug: Tacrolimus
- Sequence 3 (Active Comparator): Prograf for 1 week with full PK on Day 7, then tacrolimus Hi for 1 week with full PK on Day 14, then tacrolimus Lo for 1 week with full PK on Day 21, then Prograf with full PK on Day 28, then tacrolimus Lo for 1 week with full PK on Day 35, and then tacrolimus Hi for 1 week with full PK on Day 42
  Interventions: Drug: Prograf; Drug: Tacrolimus

INTERVENTIONS:
Drug: Prograf — Brand: Prograf Capsules, 1.0mg Tacrolimus capsules containing white to off white powder equivalent to 1.0 mg of anhydrous tacrolimus are hard gelatin capsules with white opaque body and ivory capsules.
  Other Names: Brand
Drug: Tacrolimus — Generic Hi: Generic tacrolimus Capsules, 1.0mg. Manufacturer to be determined (Aim 1).
  Other Names: Generic tacrolimus hi
Drug: Tacrolimus — Generic Lo: Generic tacrolimus Capsules, 1.0mg. Manufacturer to be determined (Aim 1).
  Other Names: Generic tacrolimus lo

SUMMARY:
The study is designed to compare the steady-state pharmacokinetics of Prograf (Brand) and the two most disparate generic formulations (Generic Hi and Generic Lo) in a fully replicated, 3-way cross-over study in stable kidney (n=36) and liver transplant (n=36) subjects.

DETAILED DESCRIPTION:
To identify the most disparate tacrolimus generic drug formulations among those currently approved in the United States. We will conduct systematic dissolution testing of the brand and all currently approved tacrolimus drug formulations using the FDA-recommended dissolution method. We propose to test and compare the 1mg capsule strength (3 production lots/ manufacturer). In addition, we will compare the different formulations in terms of potency, purity and other quality attributes. This work will be carried out in the GMP-compliant facilities of The University of Iowa Pharmaceuticals and the University of Colorado. Based on these studies the two most disparate generic tacrolimus formulations (Generic Hi and Generic Lo) will be selected and compared with the Brand (PrografR, Astellas, Deerfield, IL) in the clinical trial.

This is an open label, prospective, multicenter, randomized, replicate, six-period, three-sequence cross-over study to compare the steady state pharmacokinetics of PrografR to Generic Hi to Generic Lo in stable kidney and liver transplant subjects. The PK assessor will be blinded to the assigned treatment sequence and formulation. The person analyzing the levels and analyzing the results will be blinded to formulation sequence. Each subject will be randomized to one of the three sequences where Generic Hi and Generic Lo represent the two generics and B the brand, Prograf. The blood samples will be collected at C0 (before morning dose) and then 20, 40, 60(1hr), 80, 100, 120(2hr), 140, 160, 180(3hr) minutes, 4, 5, 6, 8 and 12 hour after dosing with each formulation. Adherence will be monitored by patient diary, pill counts, and MEMS cap. Safety and efficacy parameters will be monitored weekly.

This study will be carried out in full compliance with the rules of Good Clinical Practice (GCP) including development of an electronic database and monitoring plan.

Resulting pharmacokinetic parameters will be analyzed by a variety of pharmacokinetic tests such as narrower acceptance intervals, individual and scaled average bioequivalence was well as population pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old, male or female
2. Able to participate and willing to give written informed consent and to comply with the study visits and restrictions.
3. Subject who has received a primary or secondary kidney or liver transplant.
4. Subject who is at least 6 months post-transplant and on a stable dose of tacrolimus as defined by physician, one tacrolimus trough level within the physician defined target range within past 6 months and one additional trough level during the screening period within 30% of the physician defined target range.
5. BMI greater than or equal to 19 but less than or equal to 40.
6. Ability to perform daily finger sticks to provide blood sample

Exclusion Criteria:

1. Evidence of any acute rejection
2. Subjects who require dialysis within 6 months prior to study entry
3. Recipients of multiple organ transplants
4. Subjects who have tested positive for HBsAG or HIV, or who are recipients of organ from donors who are known to be HBsAG or HIV positive. Virology screening at the time of transplant.
5. Hep C positive subjects with liver biopsy proven recurrent disease considered relevant by physician oversight.
6. Subjects with any severe medical condition requiring acute or chronic treatment that in the investigator's opinion would interfere with study participation
7. History of malignancy, treated or untreated, with the past 2 years with the exception of carcinoma in situ or excised basal cell carcinoma, or hepatocellular carcinoma prior to transplant.
8. GFR ≤ 35 ml/min measured as estimated using the MDRD4 formula
9. Subjects with aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin ≥ 3 X upper limit of normal (ULN) or other evidence of severe liver disease
10. Subjects with white blood cell (WBC) count ≤2,000/ mm3 or with thrombocytopenia (platelet count ≤ 75,000/ mm3), with an absolute neutrophil count of ≤ 1,500/ mm3 or hemoglobin <8g/dL)
11. Subjects with clinically significant infections, requiring therapy, which, in the investigator's opinion, would interfere with the objectives of the study
12. Other mental or physical conditions which in the investigator's opinion, are considered clinically significant
13. Presence of intractable immunosuppressant complications or side effects resulting in dose adjustment of tacrolimus
14. Subjects who have been exposed to an investigational therapy within 30 days prior to enrollment or 5 half-lives of the investigational product, whichever is greater.
15. An anticipated change in the immunosuppressive regimen during subject participation other than that required by the protocol
16. Subject with severe GI disturbance or diarrhea which could interfere with tacrolimus absorption
17. Severe diabetic gastroparesis
18. Initiation of any medications that could interfere with tacrolimus blood levels, including OTC medications, herbal supplements, grapefruit or grapefruit juice.
19. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive beta human chorionic gonadotrophin (BhCG) laboratory test (> 5 mIU/mL)
20. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are

    1. women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner; women whose partners have been sterilized by vasectomy or
    2. using a highly effective method of birth control (i.e. one that results in a less than 1% per year failure rate when used consistently and correctly, such as implants, injectables, combined oral contraceptives, and some intrauterine devices (IUDs); periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) is not acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Comparison of bioequivalence between brand name prograf to generic Hi tacrolimus in all participants | Day 7, 14, 21, 28, 35, 42
  Ratio of C0, C12, AUC0-12h and Cmax and apply confidence interval (CI) testing at steady state of Prograf to generic Hi in stable kidney and liver transplant subjects
Comparison of bioequivalence between brand name prograf to generic Lo tacrolimus in all participants | Day 7, 14, 21, 28, 35, 42
  Ratio of C0, C12, AUC0-12h and Cmax and apply confidence interval (CI) testing at steady state of Prograf to Generic Lo in stable kidney and liver transplant subjects.
Comparison of bioequivalence between generic Hi tacrolimus to generic Lo tacrolimus in all participants | Day 7, 14, 21, 28, 35, 42
  Ratio of C0, C12, AUC0-12h and Cmax and apply confidence interval (CI) testing at steady state of Generic Hi to Generic Lo in stable kidney and liver transplant subjects.

SECONDARY OUTCOMES:
Comparing the bioavailability of each tacrolimus formulations in stable kidney and liver transplant subjects using the dose-normalized C0, C12, AUC0-12h and Cmax data | Day 7, 14, 21, 28, 35, 42
Evaluating intra-patient variability of tacrolimus pharmacokinetics of each formulation by comparing C0, C12, AUC0-12h, and Cmax | Day 7, 14, 21, 28, 35, 42
Evaluating and comparing the pharmacokinetics of tacrolimus metabolites in terms of C0, C12, AUC0-12h, Cmax and intra-individual variability | Day 7, 14, 21, 28, 35, 42
Comparing the safety of Prograf, Generic Hi and Generic Lo in stable kidney and liver transplant subjects | Day 7, 14, 21, 28, 35, 42
  This is a pharmacokinetic comparison study, but safety data will be collected via adverse and serious adverse event reporting as these are the standard efficacy parameters in transplant studies.
Comparing the efficacy of Prograf, Generic Hi and Generic Lo in stable kidney and liver transplant subjects | Day 7, 14, 21, 28, 35, 42
  This is a pharmacokinetic comparison study, but efficacy will be measured by kidney/liver function or biopsy-proven acute rejection or graft loss.

CONTACTS AND LOCATIONS:
Overall Officials: Rita R Alloway, PharmD, FCCP, Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio

REFERENCES:
- [Derived] Alloway RR, Vinks AA, Fukuda T, Mizuno T, King EC, Zou Y, Jiang W, Woodle ES, Tremblay S, Klawitter J, Klawitter J, Christians U. Bioequivalence between innovator and generic tacrolimus in liver and kidney transplant recipients: A randomized, crossover clinical trial. PLoS Med. 2017 Nov 14;14(11):e1002428. doi: 10.1371/journal.pmed.1002428. eCollection 2017 Nov. PMID 29135993